CLINICAL TRIAL: NCT00423137
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Evaluate the Effects of a 4-week Treatment of 15 and 30 mg b.i.d BIBW2948 BS (Inhalation Powder, Hard Capsule for HandiHaler®) on Epithelial Mucin Stores and the Safety and Efficacy in COPD Patients With Symptoms Associated With Chronic Bronchitis
Brief Title: Effect of BIBW 2948 BS in COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1219.5; 2006-001975-40
Record Dates: First submitted 2007-01-17; First posted 2007-01-18 (Estimated); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Placebo - low dose (Placebo Comparator): Twice daily (b.i.d.)
  Interventions: Drug: Placebo
- Placebo - high dose (Placebo Comparator): Twice daily (b.i.d.)
  Interventions: Drug: Placebo
- BIBW2948 - low dose (Experimental): Twice daily (b.i.d.)
  Interventions: Drug: BIBW 2948 BS
- BIBW2948 - high dose (Experimental): Twice daily (b.i.d.)
  Interventions: Drug: BIBW 2948 BS

INTERVENTIONS:
Drug: BIBW 2948 BS — Capsule
  Arms: BIBW2948 - high dose; BIBW2948 - low dose
Drug: Placebo — Capsule
  Arms: Placebo - high dose; Placebo - low dose

SUMMARY:
Study of BIBW 2948 BS in Patients with COPD and Chronic Bronchitis

ELIGIBILITY:
Inclusion Criteria:

* COPD smokers
* ages between 40 and 70

Exclusion Criteria:

* Significant other diseases
* abnormal hematology
* abnormal liver function
* psychiatric disorders
* pulmonary obstruction
* asthma, allergic rhinitis
* dependance on oxygen
* patients with history of myocardial infarction
* patients with history of cancer
* women of child bearing potential
* antiplatelet or anticoagulation therapy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-01-17 (Actual); Primary Completion 2008-07-09 (Actual); Study Completion 2008-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (6):
- United States (4):
  - 1219.5.03 Boehringer Ingelheim Investigational Site, Birmingham, Alabama
  - 1219.5.01 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1219.5.02 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1219.5.04 Boehringer Ingelheim Investigational Site, Philadelphia, Pennsylvania
- Germany (2):
  - 1219.5.06 Boehringer Ingelheim Investigational Site, Freiburg/Breisgau
  - 1219.5.05 Boehringer Ingelheim Investigational Site, Hanover

REFERENCES:
- [Derived] Woodruff PG, Wolff M, Hohlfeld JM, Krug N, Dransfield MT, Sutherland ER, Criner GJ, Kim V, Prasse A, Nivens MC, Tetzlaff K, Heilker R, Fahy JV. Safety and efficacy of an inhaled epidermal growth factor receptor inhibitor (BIBW 2948 BS) in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2010 Mar 1;181(5):438-45. doi: 10.1164/rccm.200909-1415OC. Epub 2009 Dec 10. PMID 20007923
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A randomized, double-blind, placebo-controlled, parallel group study to evaluate the effects of a 4-week treatment of 15 and 30 mg two times daily (b.i.d) BIBW2948 BS on epithelial mucin stores and the safety and efficacy in Chronic Obstructive Pulmonary (COPD) patients with symptoms associated with chronic bronchitis
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
Groups:
- Placebo 15 Milligram b.i.d: Oral inhalation of two 7.5 milligram (mg) capsules of placebo for HandiHaler® (15 mg in total) twice daily (b.i.d) over a treatment period of 4 weeks.
- Placebo 30 Milligram b.i.d: Oral inhalation of four 7.5 milligram (mg) capsules of placebo for HandiHaler® (30 mg in total) twice daily (b.i.d) over a treatment period of 4 weeks.
- BIBW2948 15 Milligram b.i.d: Oral inhalation of two 7.5 milligram (mg) capsules of BIBW2948 for HandiHaler® (15 mg in total) twice daily (b.i.d) over a treatment period of 4 weeks.
- BIBW2948 30 Milligram b.i.d: Oral inhalation of four 7.5 milligram (mg) capsules of BIBW2948 for HandiHaler® (30 mg in total) twice daily (b.i.d) over a treatment period of 4 weeks.
Period: Overall Study
Arm/Group | Placebo 15 Milligram b.i.d | Placebo 30 Milligram b.i.d | BIBW2948 15 Milligram b.i.d | BIBW2948 30 Milligram b.i.d
Started | 11 | 12 | 13 | 12
Completed | 10 | 12 | 7 | 10
Not Completed | 1 | 0 | 6 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Adverse Event Study disease worse | 1 | 0 | 3 | 1
Not completed — Adverse Event Other | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): included all treated patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo 15 Milligram b.i.d | Placebo 30 Milligram b.i.d | BIBW2948 15 Milligram b.i.d | BIBW2948 30 Milligram b.i.d | Total
Number analyzed (Participants) | 11 | 12 | 13 | 12 | 48
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.5 (7.30) | 56.4 (7.00) | 54.0 (7.99) | 59.0 (7.83) | 56.2 (7.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 7 | 3 | 16
  Male | 8 | 9 | 6 | 9 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 1 | 6
  White | 9 | 10 | 12 | 11 | 42
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Volume of Mucin Per Surface Area of Basal Lamina
Description: Change from baseline in volume of mucin per surface area of basal lamina. Volume of mucin per surface area of basal lamina (vs mu,bala) was determined by stereologic quantification of Periodic Acid Schiff's (AB/PAS) reagent staining in endobronchial biopsies at visit 2 (baseline) and at the end of the 4-week period of randomized treatment (visit 5).
Time Frame: At baseline (visit 2) and at visit 5.
Population: The treated set (TS), included all treated patients. Results are reported by pooled treatment groups (i.e. pooled group of placebo vs. pooled group of BIBW-treated patients), as defined in the statistical analysis plan.
Measure: Least Squares Mean (Standard Error); unit: micrometer^3/micrometer^2
Groups:
- Placebo Total: All patients on placebo treatment. Oral inhalation of two 7.5 milligram (mg) capsules of placebo for HandiHaler® (15 mg in total) twice daily (b.i.d) over a treatment period of 4 weeks. And oral inhalation of four 7.5 milligram (mg) capsules of placebo for HandiHaler® (30 mg in total) twice daily (b.i.d) over a treatment period of 4 weeks.
- BIBW2948 Total: All patients on BIBW2948 treatment. Oral inhalation of two 7.5 milligram (mg) capsules of BIBW2948 for HandiHaler® (15 mg in total) twice daily (b.i.d) over a treatment period of 4 weeks. And oral inhalation of four 7.5 milligram (mg) capsules of BIBW2948 for HandiHaler® (30 mg in total) twice daily (b.i.d) over a treatment period of 4 weeks.
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 23 | 25
micrometer^3/micrometer^2 | 2.565 (1.836) | 1.180 (1.676)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.5305, ANCOVA; The adjusted least squares mean is estimated based on the ANCOVA model with treatment, centre, and baseline; Difference of least square means = -1.385, Standard Error of Mean 2.181

2. Secondary Outcome: Change From Baseline of Volume of Mucin Per Volume of Epithelium (Vv mu, ep) in Endobronchial Biopsies
Description: Change from baseline of volume of mucin per volume of epithelium (Vv mu, ep) in endobronchial biopsies. The volume of mucin per volume of epithelium (Vv mu, ep), as measured by stereological quantification of AB/PAS staining in endobronchial biopsies was performed at baseline (visit 2) and at the end of the 4-week period of randomised treatment (visit 5).
Time Frame: At baseline (visit 2) and at visit 5.
Population: The treated set (TS), included all treated patients. Only patients with non-missing outcome measures were included. Results are reported by pooled treatment groups (i.e. pooled group of placebo vs. pooled group of BIBW-treated patients), as defined in the statistical analysis plan.
Measure: Least Squares Mean (Standard Error); unit: millimeter^3/millimeter^3
Groups:
- Placebo Total: All patients on Placebo Treatment. Oral inhalation of two 7.5 milligram (mg) capsules of placebo for HandiHaler® (15 mg in total) twice daily (b.i.d). And Oral inhalation of four 7.5 milligram (mg) capsules of placebo for HandiHaler® (30 mg in total) twice daily (b.i.d).
- BIBW2948 Total: All patients on BIBW2948 Treatment. Oral inhalation of two 7.5 milligram (mg) capsules of BIBW2948 for HandiHaler® (15 mg in total) twice daily (b.i.d). And Oral inhalation of four 7.5 milligram (mg) capsules of BIBW2948 for HandiHaler® (30 mg in total) twice daily (b.i.d).
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 22 | 14
millimeter^3/millimeter^3 | 0.013 (0.028) | -0.036 (0.026)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.1498, ANCOVA; The adjusted least squares mean is estimated based on the ANCOVA model with treatment, centre, and baseline; Difference of least square means = -0.049, Standard Error of Mean 0.033 — Difference to Placebo [Treatment-Placebo]

3. Secondary Outcome: Change From Baseline in Bronchoalveolar Lavage (BAL) Cell Differential (in %)
Description: Change from baseline in bronchoalveolar lavage (BAL) cell differential (in %). Differential cell counts were performed on bronchoalveolar lavage samples obtained during visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5).
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Percentage of cells
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 20 | 11
Percentage of cells
  Eosinophil [%] | 0.46 [-0.22 to 1.14] | 2.03 [0.48 to 3.58]
  Epithelial [%] | -3.22 [-10.33 to 3.89] | -0.71 [-4.70 to 3.28]
  Lymphocyte [%] | -0.15 [-0.45 to 0.15] | -0.42 [-2.14 to 1.30]
  Macrophage [%] | 2.48 [-5.38 to 10.34] | -8.68 [-26.57 to 9.21]
  Neutrophil [%] | 0.15 [-0.92 to 1.22] | 7.47 [-7.50 to 22.44]
  Squamous [%] | 0.31 [-0.32 to 0.94] | 0.40 [-0.54 to 1.34]

4. Secondary Outcome: Change From Baseline in Bronchoalveolar Lavage (BAL) Cell Count
Description: Change from baseline in bronchoalveolar lavage (BAL) cell count. Total cell counts were performed on bronchoalveolar lavage (BAL) samples obtained during visit 2 (baseline) and at the end of the 4-week period of randomised treatment.
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: Cells per milliliter
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 20 | 11
Cells per milliliter
  Eosinophil | 0.001 [-0.001 to 0.003] | 0.005 [-0.000 to 0.010]
  Epithelial | -0.001 [-0.008 to 0.006] | -0.007 [-0.026 to 0.012]
  Lymphocyte | -0.001 [-0.002 to 0.001] | 0.001 [-0.004 to 0.005]
  Macrophage | 0.016 [-0.188 to 0.220] | -0.206 [-0.446 to 0.034]
  Neutrophil | -0.001 [-0.005 to 0.003] | 0.004 [-0.021 to 0.028]
  Squamous | 0.000 [-0.000 to 0.001] | 0.000 [-0.001 to 0.002]

5. Secondary Outcome: Change From Baseline in Log MUC2 Mucin Gene Expression (RNA) Obtained in Epithelial Brushings
Description: Change from baseline in log MUC2 Mucin gene expression (RNA) obtained in epithelial brushings. Gene expression levels of the gel-forming mucins (MUC2) were quantified using two-step real time polymerase chain reaction (PCR) from RNA extracted from the cells obtained from the epithelial brushings during the endobronchial biopsy at visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5).
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Log (fold change)
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 20 | 12
Log (fold change) | 0.076 (0.343) | 0.411 (0.325)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.4472, ANCOVA; The adjusted least squares mean is estimated based on the ANCOVA model with treatment, centre, and baseline; Difference of least square means = 0.335, Standard Error of Mean 0.434 — Difference to Placebo [Treatment-Placebo]

6. Secondary Outcome: Change From Baseline in Log Mucin Gene (MUC5AC) Expression Level Obtained in Epithelial Brushings
Description: Change from baseline in log mucin gene (MUC5AC) expression level obtained in epithelial brushings. Gene expression levels of the gel-forming mucins (MUC5AC) were quantified using two-step real time polymerase chain reaction (PCR) from RNA extracted from the cells obtained from the epithelial brushings during the endobronchial biopsy at visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5).
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Log (fold change)
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 20 | 12
Log (fold change) | 0.074 (0.275) | -0.067 (0.247)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.6829, ANCOVA; The adjusted least squares mean is estimated based on the ANCOVA model with treatment, centre, and baseline; Difference of least square means = -0.141, Standard Error of Mean 0.342 — Difference to Placebo [Treatment-Placebo]

7. Secondary Outcome: Change From Baseline in Log Mucin Gene (MUC5B) Expression Level Obtained in Epithelial Brushings
Description: Change from baseline in log mucin gene (MUC5B) expression level obtained in epithelial brushings.
  Gene expression levels of the gel-forming mucins (MUC5B) were quantified using two-step real time polymerase chain reaction (PCR) from RNA extracted from the cells obtained from the epithelial brushings during the endobronchial biopsy at visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5).
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Log (fold change)
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 20 | 12
Log (fold change) | -0.377 (0.309) | 0.194 (0.296)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.1565, ANCOVA; The adjusted least squares mean is estimated based on the ANCOVA model with treatment, centre, and baseline; Difference of least square means = 0.571, Standard Error of Mean 0.391 — Difference to Placebo [Treatment-Placebo]

8. Secondary Outcome: Change From Baseline in Log Mucin Gene (MUC8) Expression Level Obtained in Epithelial Brushings
Description: Change from baseline in log mucin gene (MUC8) expression level obtained in epithelial brushings. Gene expression levels of the gel-forming mucins (MUC8) were quantified using two-step real time polymerase chain reaction (PCR) from RNA extracted from the cells obtained from the epithelial brushings during the endobronchial biopsy at visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5).
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Log (fold change)
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 20 | 12
Log (fold change) | 0.639 (0.961) | 1.720 (0.865)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.3709, ANCOVA; The adjusted least squares mean is estimated based on the ANCOVA model with treatment, centre, and baseline; Difference of least square means = 1.081, Standard Error of Mean 1.185 — Difference to Placebo [Treatment-Placebo]

9. Secondary Outcome: Change From Baseline in Epidermal Growth Factor Receptor (EGRF) Internalization Assay in Epithelial Brushings - Cells With Bright Spots With Marker
Description: Change in percentage of cells with bright spots with marker. The degree of EGFR internalization (and hence activation) was measured using antibody or ligand labeling techniques in epithelial brushing samples obtained during the endobronchial biopsy at visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5). Measurements visit 2 are used to standardize measurements at visit 5, and the standardized visit 5 value is calculated in percent (%) control as (visit5/visit2*100).
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of baseline level
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 16 | 9
Percentage of baseline level | 103.122 (9.889) | 51.039 (13.19)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.0044, ANCOVA; The adjusted least squares mean is estimated based on the one way ANOVA model with Treatment; Difference of least square means = -52.083, Standard Error of Mean 16.48 — Difference to Placebo [Treatment-Placebo]

10. Secondary Outcome: Change From Baseline in Epidermal Growth Factor Receptor (EGRF) Internalization Assay in Epithelial Brushings - EGRF Spots at Nucleus
Description: Change in number of EGRF spots at nucleus. The degree of EGFR internalization (and hence activation) was measured using antibody or ligand labeling techniques in epithelial brushing samples obtained during the endobronchial biopsy at visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5). Measurements visit 2 are used to standardize measurements at visit 5, and the standardized visit 5 value is calculated in percent (%) control as (visit5/visit2*100).
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of baseline level
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 16 | 9
Percentage of baseline level | 112.955 (13.15) | 45.943 (17.53)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.0056, ANCOVA; The adjusted least squares mean is estimated based on the one way ANOVA model with Treatment; Difference of least square means = -67.012, Standard Error of Mean 21.29 — Difference to Placebo [Treatment-Placebo]

11. Secondary Outcome: Change From Baseline in Epidermal Growth Factor Receptor (EGFR) Internalization Assay in Epithelial Brushings - EGRF Spots With Marker
Description: Change in number of EGRF spots with marker per cell. The degree of EGFR internalization (and hence activation) was measured using antibody or ligand labeling techniques in epithelial brushing samples obtained during the endobronchial biopsy at visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5). Measurements visit 2 are used to standardize measurements at visit 5, and the standardized visit 5 value is calculated in percent (%) control as (visit5/visit2*100).
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of baseline level
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 16 | 9
Percentage of baseline level | 106.671 (11.05) | 44.100 (14.74)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.0025, ANCOVA; The adjusted least squares mean is estimated based on the one way ANOVA model with Treatment; Difference of least square means = -62.571, Standard Error of Mean 18.42 — Difference to Placebo [Treatment-Placebo]

12. Secondary Outcome: Change From Baseline in Epidermal Growth Factor Receptor (EGFR) Internalization Assay in Epithelial Brushings - Total Area Bright Spots With Marker
Description: Change in total area bright spots with marker. The degree of EGFR internalization (and hence activation) was measured using antibody or ligand labeling techniques in epithelial brushing samples obtained during the endobronchial biopsy at visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5). Measurements visit 2 are used to standardize measurements at visit 5, and the standardized visit 5 value is calculated in percent (%) control as (visit5/visit2*100).
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of baseline level
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 16 | 9
Percentage of baseline level | 95.397 (11.28) | 55.330 (15.04)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.0439, ANCOVA; The adjusted least squares mean is estimated based on the one way ANOVA model with Treatment; Difference of least square means = -40.067, Standard Error of Mean 18.80 — Difference to Placebo [Treatment-Placebo]

13. Secondary Outcome: Change From Baseline in Epidermal Growth Factor Receptor (EGFR) Internalization Assay in Epithelial Brushings - EGFR Spots
Description: Change in number of EGFR spots per cell. The degree of EGFR internalization (and hence activation) was measured using antibody or ligand labeling techniques in epithelial brushing samples obtained during the endobronchial biopsy at visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5). Measurements visit 2 are used to standardize measurements at visit 5, and the standardized visit 5 value is calculated in % control as (visit5/visit2*100).
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of baseline level
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 16 | 9
Percentage of baseline level | 117.074 (12.78) | 59.614 (17.04)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.0129, ANCOVA; The adjusted least squares mean is estimated based on the one way ANOVA model with Treatment; Difference of least square means = -57.460, Standard Error of Mean 21.30 — Difference to Placebo [Treatment-Placebo]

14. Secondary Outcome: Change From Baseline in Epidermal Growth Factor Receptor (EGFR) Internalization Assay in Epithelial Brushings - EGFR Spots at Nucleus With Marker
Description: Change in number of EGFR spots at nucleus per cell with marker. The degree of EGFR internalization (and hence activation) was measured using antibody or ligand labeling techniques in epithelial brushing samples obtained during the endobronchial biopsy at visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5). Measurements visit 2 are used to standardize measurements at visit 5, and the standardized visit 5 value is calculated in % control as (visit5/visit2*100).
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Percentage of baseline level
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 16 | 9
Percentage of baseline level | 110.045 (10.27) | 54.713 (13.69)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.0037, ANCOVA; The adjusted least squares mean is estimated based on the one way ANOVA model with Treatment; Difference of least square means = -55.332, Standard Error of Mean 17.11 — Difference to Placebo [Treatment-Placebo]

15. Secondary Outcome: Change From Baseline in Number of Goblet Cells Per Surface Area of Basel Lamina
Description: Change from baseline in number of goblet cells per surface area of basel lamina, using endobronchial biopsies, taken at visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5).
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: cells/micrometer^2
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 21 | 11
cells/micrometer^2 | 0.001 (0.0008) | 0.001 (0.0008)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.9076, ANCOVA; The adjusted least squares mean is estimated based on the ANCOVA model with treatment, centre, and baseline; Difference of least square means = -0.0000, Standard Error of Mean 0.0010 — Difference to Placebo [Treatment-Placebo]

16. Secondary Outcome: Change From Baseline in Number of Goblet Cells Per Volume of Epithelium
Description: Change from baseline in number of goblet cells per volume of epithelium, using endobronchial biopsies, taken at visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5).
Time Frame: At baseline (visit 2) and visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Cells/micrometer^3
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 21 | 11
Cells/micrometer^3 | 14332.8 (12812) | 879.408 (12583)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.4121, ANCOVA; The adjusted least squares mean is estimated based on the ANCOVA model with treatment, centre, and baseline; Difference of least square means = -13453, Standard Error of Mean 16118 — Difference to Placebo [Treatment-Placebo]

17. Secondary Outcome: Change From Baseline in Goblet Cell Volume
Description: Change from baseline in goblet cell volume, using endobronchial biopsies, taken at visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5).
Time Frame: At baseline (visit 2) and visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: micrometer^3
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 21 | 11
micrometer^3 | -607.26 (239.71) | -685.87 (236.65)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.7948, ANCOVA; The adjusted least squares mean is estimated based on the ANCOVA model with treatment, centre, and baseline; Difference of least square means = -78.619, Standard Error of Mean 298.91 — Difference to Placebo [Treatment-Placebo]

18. Secondary Outcome: Change From Baseline of Interleukin-8 (IL-8) Levels in Bronchoalveolar Lavage
Description: Change from baseline of Interleukin-8 (IL-8) levels in bronchoalveolar lavage. IL-8 levels, were measured by enzyme linked immunosorbent assay in bronchoalveolar lavage samples at visit 2 (baseline) and at the end of the 4-week period of treatment (visit 5).
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nanogram per milliliter
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 21 | 12
nanogram per milliliter | -0.069 (0.070) | 0.126 (0.077)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.0640, ANCOVA; The adjusted least squares mean is estimated based on the ANCOVA model with treatment, centre, and baseline; Difference of least square means = 0.195, Standard Error of Mean 0.101 — Difference to Placebo [Treatment-Placebo]

19. Secondary Outcome: Change From Baseline in Myeloperoxidase (MPO) Levels in Bronchoalveolar Lavage
Description: Change from baseline in Myeloperoxidase (MPO) levels in bronchoalveolar lavage. Myeloperoxidase (MPO) activity levels were measured by enzyme linked immunosorbent or radioimmunoassay assay in bronchoalveolar lavage samples at visit 2 (baseline) and at the end of the 4-week period of randomised treatment (visit 5).
Time Frame: At baseline (visit 2) and at visit 5.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: microgram per deciliter
Arm/Group | Placebo Total | BIBW2948 Total
Number analyzed (Participants) | 21 | 12
microgram per deciliter | -0.003 (0.003) | 0.005 (0.003)
Statistical Analysis 1: Comparison: Placebo Total vs BIBW2948 Total; Test type: Other; p = 0.0587, ANCOVA; The adjusted least squares mean is estimated based on the ANCOVA model with treatment, centre, and baseline; Difference of least square means = 0.007, Standard Error of Mean 0.004 — Difference to Placebo [Treatment-Placebo]

ADVERSE EVENTS:
Time Frame: From first drug intake until last drug intake + 14 days, up to 4 weeks + 14 days.
Description: The treated set (TS), included all treated patients.
Groups:
- Total: All patients in the study combined. (Placebo + BIBW2948)
Arm/Group | Placebo 15 Milligram b.i.d | Placebo 30 Milligram b.i.d | Placebo Total | BIBW2948 15 Milligram b.i.d | BIBW2948 30 Milligram b.i.d | BIBW2948 Total | Total
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/23 | 0/13 | 0/12 | 0/25 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/23 | 3/13 | 1/12 | 4/25 | 4/48
Other Adverse Events (participants affected / at risk) | 9/11 | 9/12 | 18/23 | 11/13 | 9/12 | 20/25 | 38/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo 15 Milligram b.i.d (N=11) | Placebo 30 Milligram b.i.d (N=12) | Placebo Total (N=23) | BIBW2948 15 Milligram b.i.d (N=13) | BIBW2948 30 Milligram b.i.d (N=12) | BIBW2948 Total (N=25) | Total (N=48)
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo 15 Milligram b.i.d (N=11) | Placebo 30 Milligram b.i.d (N=12) | Placebo Total (N=23) | BIBW2948 15 Milligram b.i.d (N=13) | BIBW2948 30 Milligram b.i.d (N=12) | BIBW2948 Total (N=25) | Total (N=48)
Bundle branch block right (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Chest pain (General disorders) | 2 | 1 | 3 | 0 | 0 | 0 | 3
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Influenza like illness (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Oedema peripheral (General disorders) | 2 | 0 | 2 | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 1 | 0 | 1 | 2 | 1 | 3 | 4
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hordeolum (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 2 | 0 | 2 | 4
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 2 | 0 | 2 | 2
Pulmonary function test decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 2
Headache (Nervous system disorders) | 0 | 3 | 3 | 2 | 2 | 4 | 7
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Sinus headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 6 | 4 | 2 | 6 | 12
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 1 | 1 | 2 | 5
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 3 | 0 | 3 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 2
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 0 | 0 | 0 | 4
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.